CLINICAL TRIAL: NCT01421511
Title: A Phase 3 Randomized, Double-Blind, Multicenter Study Comparing the Efficacy and Safety of IV to Oral 6-Day TR-701 Free Acid and IV to Oral 10-Day Linezolid for the Treatment of ABSSSI
Brief Title: TR-701 FA vs Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1986-010; TR701-113 (Other: TriusRX Unique ID)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections
Keywords: ABSSSI; Tedizolid Phosphate; TR-701; Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TR-701 FA (Experimental): • TR-701 FA IV followed by TR-701 FA tablets
  Interventions: Drug: TR-701 FA
- Linezolid (Active Comparator): • Linezolid IV followed by Linezolid Tablets
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: TR-701 FA — * TR-701 FA 200 mg once daily in 250 mL sterile saline for injection as a 60 minute IV infusion
  * TR-701 FA Tablets, 200 mg, orally once daily
  Arms: TR-701 FA
Drug: Linezolid — * Linezolid 600 mg IV Injection twice daily in 300 mL sterile saline for injection as a 60 minute IV infusion
  * Linezolid Tablets, 600 mg, orally every 12 hours
  Arms: Linezolid

SUMMARY:
This is a randomized, double-blind, double-dummy, multicenter, global Phase 3 study of IV to oral TR-701 FA 200 mg once daily for 6 days versus IV to oral Zyvox® (linezolid) 600 mg every 12 hours for 10 days for the treatment of ABSSSI in adults. Patients are to start treatment with at least 2 IV doses and may receive IV therapy for the entire treatment duration.

Approximately 100 to 140 sites globally will participate in this study. Patients with an ABSSSI caused by suspected or documented gram positive pathogen(s) at baseline will be randomized 1:1 to study treatment.

DETAILED DESCRIPTION:
The primary objective is to determine the noninferiority (NI) in the early clinical response rate of intravenous (IV) to oral 6 day TR-701 free acid (FA) compared with that of IV to oral 10-day linezolid treatment at 48-72 hours after the first infusion of study drug in the intent-to-treat (ITT) analysis set in patients with acute bacterial skin and skin structure infections (ABSSSI).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring IV antibiotic therapy and with systemic signs of infection diagnosed with ABSSSI.
* Diagnosed with Cellulitis/ erysipelas, major cutaneous abscess, or wound infections

Exclusion Criteria:

* Uncomplicated skin infections
* Severe sepsis or septic shock
* ABSSSI solely due to gram-negative pathogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2013-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Director — Trius Therapeutics
Locations (116):
- United States (35):
  - Trius investigator site 159, Dothan, Alabama
  - Trius investigator site 103, Chula Vista, California
  - Trius investigator site 143, Escondido, California
  - Trius investigator site 105, La Mesa, California
  - Trius investigator site 106, Long Beach, California
  - Trius investigator site 157, Long Beach, California
  - Trius investigator site 142, National City, California
  - Trius investigator site 170, San Diego, California
  - Trius investigator site 167, Santa Ana, California
  - Trius investigator site 168, Stockton, California
  - Trius investigator site 141, Sylmar, California
  - Trius investigator site 139, Denver, Colorado
  - Trius investigator site 137, Newark, Delaware
  - Trius investigator site 166, Edgewater, Florida
  - Trius investigator site 101, Columbus, Georgia
  - Trius investigator site 138, Carmel, Indiana
  - Trius investigator site 144, Owensboro, Kentucky
  - Trius investigator site 150, Baton Rouge, Louisiana
  - Trius investigator site 165, Eunice, Louisiana
  - Trius investigator site 154, Boston, Massachusetts
  - Trius investigator site 146, Springfield, Massachusetts
  - Trius investigator site 136, West Roxbury, Massachusetts
  - Trius investigator site 163, Royal Oak, Michigan
  - Trius investigator site 153, Minneapolis, Minnesota
  - Trius investigator site 149, Picayune, Mississippi
  - Trius investigator site 164, Creve Coeur, Missouri
  - Trius investigator site 160, Las Vegas, Nevada
  - Trius investigator site 147, Teaneck, New Jersey
  - Trius investigator site 140, Columbus, Ohio
  - Trius investigator site 162, Lima, Ohio
  - Trius investigator site 161, Rapid City, South Dakota
  - Trius investigator site 155, Franklin, Tennessee
  - Trius investigator site 145, Memphis, Tennessee
  - Trius investigator site 169, Smyrna, Tennessee
  - Trius investigator site 148, Houston, Texas
- Argentina (11):
  - Trius investigator site 352, Cludadela, Buenos Aires
  - Trius investigator site 354, General Roriquez, Buenos Aires
  - Trius investigator site 350, La Plata, Buenos Aires
  - Trius investigator site 353, Luján, Buenos Aires
  - Trius investigator site 354, Buenos Aires
  - Trius investigator site 355, Buenos Aires
  - Trius investigator site 351, Cludad Autonoma de Buenos Aires
  - Trius investigator site 358, La Plata
  - Trius investigator site 357, Mar del Plata
  - Trius investigator site 359, Paraná, Entre Rios
  - Trius investigator site 356, Rosario
- Australia (7):
  - Trius investigator 500, Cairns, Queensland
  - Trius investigator 501, Herston, Queensland
  - Trius investigator 503, Nambour, Queensland
  - Trius investigator 506, Southport, Queensland
  - Trius investigator 502, Woolloongabba, Queensland
  - Trius investigator 504, Woolloongabba, Queensland
  - Trius investigator 505, Richmond, Victoria
- Brazil (14):
  - Trius investigator site 362, Belo Horizonte, MG, Brazil
  - Trius investigator site 361, Belo Horizonte, MG, Brazil
  - Trius investigator site 363, Porto Alegre, RS, Brazil
  - Trius investigator site 364, Campinas, SP, Brazil
  - Trius investigator site 361, Belo Horizonte
  - Trius investigator site 362, Belo Horizonte
  - Trius investigator site 365, Belo Horizonte
  - Trius investigator site 364, Campinas
  - Trius investigator site 366, Curitiba
  - Trius investigator site 367, Curitiba
  - Trius investigator site 369, Jaú
  - Trius investigator site 363, Porto Alegre
  - Trius investigator site 370, Porto Alegre
  - Trius investigator site 360, São Paulo
- Germany (5):
  - Trius investigator site 208, Dresden, Saxony
  - Trius investigator site 206, Quedlinburg, Saxony-Anhalt
  - Trius investigator site 204, Lübeck, Schleswig-Holstein
  - Trius investigator site 207, Berlin
  - Trius investigator site 205, Hamburg
- Mexico (4):
  - Trius investigator site 380, Guadalajara
  - Trius investigator site 381, Guadalajara
  - Trius investigator site 382, Mexico City
  - Trius investigator site 383, Monterrey
- New Zealand (2):
  - Trius investigator 521, Otahuhu, Auckland
  - Trius investigator 520, Sydenham, Christchurch
- Poland (6):
  - Trius investigator site 216, Bydgoszcz
  - Trius investigator site 211, Lodz
  - Trius investigator site 214, Lublin
  - Trius investigator site 213, Poznan
  - Trius investigator site 215, Szczecin
  - Trius investigator site 212, Warsaw
- Russia (14):
  - Trius investigator site 292, Vsevolozhsk, Leningradskaya Oblast'
  - Trius investigator site 287, Barmaul
  - Trius investigator site 286, Irkutsk
  - Trius investigator site 293, Lipetsk
  - Trius investigator site 295, Moscow
  - Trius investigator site 290, Moscow
  - Trius investigator site 291, Moscow
  - Trius investigator site 288, Moscow
  - Trius investigator site 297, Novosibirsk
  - Trius investigator site 285, Novosibirsk
  - Trius investigator site 294, Saint Petersburg
  - Trius investigator site 289, Saint Petersburg
  - Trius investigator site 296, Saint Petersburg
  - Trius investigator site 298, Tomsk
- South Africa (12):
  - Trius investigator 444, Worscester, Cape
  - Trius investigator 443, Port Elizabeth, Eastern Cape
  - Trius investigator site 442, Bloemfontein, Free States
  - Trius investigator site 441, Blowmfontein, Free States
  - Trius investigator 451, Centurion, Gauteng
  - Trius investigator site 440, Gezina Pretoria, Gauteng
  - Trius investigator 450, Pretoria, Gauteng
  - Trius investigator 449, Pretoria, Gauteng
  - Trius investigator 448, Dundee, KwaZulu-Natal
  - Trius investigator 446, Middelburg, Mpumalanga
  - Trius investigator 447, Breyten, Mpunalanga
  - Trius investigator site 445, Benoni
- Spain (6):
  - Trius investigator site 273, Mataró, Barcelona
  - Trius investigator site 272, Alcorcón, Madrid
  - Trius investigator site 275, Majadahonda, Madrid
  - Trius investigator site 277, Barakaldo, Vizcaya
  - Trius investigator site 276, Madrid
  - Trius investigator site 274, Santander

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sandison T, De Anda C, Fang E, Das AF, Prokocimer P. Clinical Response of Tedizolid versus Linezolid in Acute Bacterial Skin and Skin Structure Infections by Severity Measure Using a Pooled Analysis from Two Phase 3 Double-Blind Trials. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02687-16. doi: 10.1128/AAC.02687-16. Print 2017 May. PMID 28264845
- [Derived] Nathwani D, Corey R, Das AF, Sandison T, De Anda C, Prokocimer P. Early Clinical Response as a Predictor of Late Treatment Success in Patients With Acute Bacterial Skin and Skin Structure Infections: Retrospective Analysis of 2 Randomized Controlled Trials. Clin Infect Dis. 2017 Jan 15;64(2):214-217. doi: 10.1093/cid/ciw750. Epub 2016 Dec 21. PMID 28003218
- [Derived] Powers JH 3rd, Das AF, De Anda C, Prokocimer P. Clinician-reported lesion measurements in skin infection trials: Definitions, reliability, and association with patient-reported pain. Contemp Clin Trials. 2016 Sep;50:265-72. doi: 10.1016/j.cct.2016.08.010. Epub 2016 Aug 13. PMID 27530088
- [Derived] Shorr AF, Lodise TP, Corey GR, De Anda C, Fang E, Das AF, Prokocimer P. Analysis of the phase 3 ESTABLISH trials of tedizolid versus linezolid in acute bacterial skin and skin structure infections. Antimicrob Agents Chemother. 2015 Feb;59(2):864-71. doi: 10.1128/AAC.03688-14. Epub 2014 Nov 24. PMID 25421472
- [Derived] Lodise TP, Fang E, Minassian SL, Prokocimer PG. Platelet profile in patients with acute bacterial skin and skin structure infections receiving tedizolid or linezolid: findings from the Phase 3 ESTABLISH clinical trials. Antimicrob Agents Chemother. 2014 Dec;58(12):7198-204. doi: 10.1128/AAC.03509-14. Epub 2014 Sep 22. PMID 25246392
- [Derived] Moran GJ, Fang E, Corey GR, Das AF, De Anda C, Prokocimer P. Tedizolid for 6 days versus linezolid for 10 days for acute bacterial skin and skin-structure infections (ESTABLISH-2): a randomised, double-blind, phase 3, non-inferiority trial. Lancet Infect Dis. 2014 Aug;14(8):696-705. doi: 10.1016/S1473-3099(14)70737-6. Epub 2014 Jun 5. PMID 24909499

RESULTS

PARTICIPANT FLOW:
Groups:
- Tedizolid Phosphate: IV to oral tedizolid phosphate 200 mg once daily for 6 days followed by 4 days of placebo.
- Linezolid: IV to oral linezolid 600 mg twice daily for 10 days.
Period: Overall Study
Arm/Group | Tedizolid Phosphate | Linezolid
Started | 332 | 334
Completed | 313 | 306
Not Completed | 19 | 28
Not completed — Lost to Follow-up | 11 | 14
Not completed — Randomized but didn't receive study drug | 1 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Tedizolid Phosphate: IV to oral tedizolid phosphate 200 mg once daily for six days followed by four days of placebo.
- Total: Total of all reporting groups
Arm/Group | Tedizolid Phosphate | Linezolid | Total
Number analyzed (Participants) | 332 | 334 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (15.79) | 45.6 (15.57) | 45.6 (15.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 120 | 227
  Male | 225 | 214 | 439

OUTCOME MEASURES:

1. Primary Outcome: The Early Clinical Response Rate
Description: Responder: No increase in lesion surface area from baseline.
Time Frame: 48-72 hours
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
participants | 283 | 276
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the early clinical response rates at 48 to 72 Hours after the first infusion of study drug using the method of Miettinen and Nurminen without stratification. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10%; Risk Difference (RD) = 2.6, 95% CI 2-sided [-3.0 to 8.2] — Risk difference corresponds to the tedizolid responder rate minus the linezolid responder rate

2. Secondary Outcome: Clinical Response at the End of Therapy Visit
Description: Responder: No increase in lesion surface area from baseline.
Time Frame: Day 11
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
participants | 289 | 294
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the programmatic clinical response at the EOT visit using the method of Miettinen and Nurminen without stratification. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Hierarchical testing procedure of Westfall and Krishen used to control for inflation of the overall type I error rate. If NI is declared for the primary, NI will be tested for the secondary outcomes in this order: Secondary Outcomes Measures 2 to 5; Risk Difference (RD) = -1.0, 95% CI 2-sided [-6.1 to 4.1] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

3. Secondary Outcome: Clinical Response at the End of Therapy Visit in the Clinically Evaluable at End of Therapy Analysis Set
Description: Responder: No increase in lesion surface area from baseline.
Time Frame: End of Therapy Day 11
Population: All randomized participants receiving minimal study therapy, completed EOT assessment, no concomitant systemic antibiotic therapy and no confounding events or factors.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 304 | 299
participants | 272 | 280
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the Investigator's assessment of clinical response at the EOT Visit using the method of Miettinen and Nurminen without stratification. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Risk Difference (RD) = -4.1, 95% CI 2-sided [-8.8 to 0.3] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

4. Secondary Outcome: Investigator's Assessment of Clinical Success at the Post Treatment Evaluation Visit
Description: Clinical success defined as resolution/near resolution of disease specific signs and symptoms, absence/near resolution of baseline systemic signs of infection, and no further antibiotic therapy required for treatment of primary ABSSSI lesion.
Time Frame: Post-Treatment Evaluation (7-14 days after the End of Therapy)
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
participants | 292 | 293
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the clinical success rate based on the Investigator's assessment of clinical response at the PTE Visit using the method of Miettinen and Nurminen without stratification. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Risk Difference (RD) = 0.3, 95% CI 2-sided [-4.8 to 5.3] — Risk difference corresponds to the tedizolid clinical success rate minus the linezolid clinical success rate

5. Secondary Outcome: Investigator's Assessment of Clinical Success of the Post Therapy Evaluation Visit in Clinically Evaluable-Post Treatment Evaluation Analysis Set.
Description: Clinical success defined as resolution/near resolution of disease specific signs and symptoms, absence/near resolution of baseline systemic signs of infection, no new signs, symptoms or complications attributable to the ABSSSI and no further antibiotic therapy required for treatment of primary ABSSSI lesion.
Time Frame: Post-Treatment Evaluation (7-14 days after the End of Therapy)
Population: All randomized participants receiving minimal study therapy, completed EOT and PTE Investigator's assessments, no concomitant systemic antibiotic therapy through PTE, and no confounding events or factors.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 290 | 280
participants | 268 | 269
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Risk Difference (RD) = -3.7, 95% CI 2-sided [-7.7 to 0.2] — Risk difference corresponds to the tedizolid clinical success rate minus the linezolid clinical success rate

6. Secondary Outcome: Investigator's Assessment of Clinical Response at the 48-72 Hour Visit
Description: Clinical improvement defined as improvement in overall clinical status.
Time Frame: 48-72 Hours
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
participants | 304 | 302
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the Investigator's assessment of clinical response at the 48-72 Hour Visit using the method of Miettinen and Nurminen without stratification; Test type: Superiority or Other; Risk Difference (RD) = 1.2, 95% CI 2-sided [-3.3 to 5.6] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

7. Secondary Outcome: Investigator's Assessment of Clinical Response at the Day-7 Visit
Description: Clinical improvement defined as improvement in overall clinical status.
Time Frame: Day 7
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
participants | 309 | 308
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the Investigator's assessment of clinical response at the Day 7 Visit using the method of Miettinen and Nurminen without stratification; Test type: Superiority or Other; Risk Difference (RD) = 0.9, 95% CI 2-sided [-3.2 to 4.9] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

8. Secondary Outcome: Change From Baseline in Patient-reported Pain, by Study Visit
Description: 0=no pain, 10=worst pain Only 1 visit per participant for Day 4-6, only 1 visit for Day 7-9, and only 1 visit for Day 10-13.
Time Frame: Multiple
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 334
units on a scale
  Day 2 | -1.7 (2.05) | -2.1 (2.29)
  Day 4-6 | -3.1 (2.67) | -3.3 (2.56)
  Day 7-9 | -4.9 (2.89) | -4.9 (2.96)
  Day 10-13 | -5.4 (2.80) | -5.6 (2.84)

ADVERSE EVENTS:
Time Frame: Collected from signing of the ICF through the late follow-up visit (up to 38 days).
Description: Numbers for at risk include all treated participants.
Arm/Group | Tedizolid Phosphate | Linezolid
Serious Adverse Events (participants affected / at risk) | 7/331 | 9/327
Other Adverse Events (participants affected / at risk) | 84/331 | 90/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (N=331) | Linezolid (N=327)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Cellutitis (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphyloccal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (N=331) | Linezolid (N=327)
Diarrhoea (Gastrointestinal disorders) | 11 | 17
Nausea (Gastrointestinal disorders) | 26 | 36
Vomiting (Gastrointestinal disorders) | 10 | 17
Fatigue (General disorders) | 8 | 7
Abscess (Infections and infestations) | 14 | 10
Cellulitis (Infections and infestations) | 9 | 6
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 7
Dizziness (Nervous system disorders) | 4 | 7
Headache (Nervous system disorders) | 20 | 22

LIMITATIONS AND CAVEATS:
Analyses for this study were conducted using 2 statistical plans, 1 for the US FDA and 1 for the EMA, to address differing guidance on the development of antibacterials. These differences are reflected in the EudraCT and clinicaltrials.gov records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to pursue publication of the results of the study in cooperation with a lead Investigator, subject to the terms and conditions of the clinical study agreement between the Sponsor and Investigators. Sponsor approval in writing is required for publication of any data subsets. Final authorship will be determined in accordance with the International Committee of Medical Journal Editors definition of authorship.